CLINICAL TRIAL: NCT03083821
Title: A Clinical Study to Evaluate the Steady State Pharmacokinetics of Baraclude in Participants With Hepatitis B Virus Infection
Brief Title: A Study to Provide a Better Understanding of Baraclude's Pharmacokinetic Properties in a Real World Clinical Setting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI463-528
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-02

CONDITIONS: Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: Baraclude

INTERVENTIONS:
Drug: Baraclude — Specified dose on specified day

SUMMARY:
A Pharmacokinetics study of Baraclude in a real world clinical setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

* Participants with chronic hepatitis B (CHB) (excluding participants with a superinfection) who have been confirmed to have CHB.
* Participants who are being treated with 0.5 mg daily Baraclude for a minimum of 10 consecutive days prior to the study enrollment.
* Body mass index (BMI) of 18.5 to 30 kg/m2 (BMI = body weight [kg]/height [m]2)

Exclusion Criteria:

* Current or recent (within 3 months of Baraclude administration) gastrointestinal disease that could impact upon the absorption of study drug.
* Any gastrointestinal surgery that could impact upon the absorption of study drug.
* Donation of blood to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration (within 2 weeks for plasma only).

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hachioji-shi, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Baraclude: Baraclude, 0.5 mg, 1 dose at 9:00 am of Day 1 (+/- 30 minutes), oral
Period: Overall Study
Arm/Group | Baraclude
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Baraclude
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All Treated Participants
  Years | 55.0 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax is defined as the peak plasma concentration
Time Frame: Up to 24 hours
Population: All treated participants with available pharmacokinetics data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baraclude
Number analyzed (Participants) | 6
ng/mL | 8.17 (2.517)

2. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax)
Description: Tmax is defined as the time of maximum observed plasma concentration, measured in hours
Time Frame: Up to 24 hours
Population: All treated participants with available pharmacokinetics data
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Baraclude
Number analyzed (Participants) | 6
Hours | 0.667 (0.2582)

3. Primary Outcome: Trough Observed Plasma (Predose) Concentration (Ctrough)
Description: Ctrough is defined as the trough in observed plasma (predose) concentrations
Time Frame: prior to administration of drug (predose)
Population: All treated participants with available pharmacokinetics data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baraclude
Number analyzed (Participants) | 6
ng/mL | 0 (0)

4. Primary Outcome: Observed Plasma Concentration at 24 Hours Postdose (C24)
Description: C24 is defined as the observed plasma concentration at 24 hours post-dose
Time Frame: 24 hours post-dose
Population: All treated participants with available pharmacokinetics data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baraclude
Number analyzed (Participants) | 6
ng/mL | 0.435 (0.0678)

5. Primary Outcome: Area Under the Concentration-time Curve in One Dosing Interval [AUC(TAU)]
Description: AUC(TAU) is defined as the area under the concentration-time curve in one dosing interval
Time Frame: Up to 24 hours
Population: All treated participants with available pharmacokinetics data
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Baraclude
Number analyzed (Participants) | 6
h*ng/mL | 21.8 (4.53)

6. Primary Outcome: Apparent Total Body Clearance (CLT/F)
Description: CLT/F is defined as the apparent total body clearance
Time Frame: Up to 24 hours
Population: All treated participants with available pharmacokinetics data
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Baraclude
Number analyzed (Participants) | 6
mL/min | 397 (81.7)

ADVERSE EVENTS:
Time Frame: AE information should begin at initiation of study treatment until 100 days after discontinuation
Arm/Group | Baraclude
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submitter for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT03083821/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT03083821/SAP_001.pdf